CLINICAL TRIAL: NCT03602261
Title: A Multi-Center, Randomized, Two-Cohort Phase 2 Study to Evaluate the Safety, Efficacy, Pharmacokinetics and Pharmacodynamics of CTAP101 (Calcifediol) Extended-Release Capsules to Treat Secondary Hyperparathyroidism in Subjects With Vitamin D Insufficiency and Chronic Kidney Disease Requiring Regular Hemodialysis.
Brief Title: Safety, Efficacy, PK and PD of CTAP101 (Calcifediol) ER Capsules for SHPT in HD Patients VDI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Cohort 1 completed and cohort 2 terminated prior to initiation per company decision
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTAP101-CL-2010
Record Dates: First submitted 2018-07-13; First posted 2018-07-26 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Secondary Hyperparathyroidism Due to Renal Causes; Chronic Kidney Diseases; Vitamin D Deficiency; Stage 5 Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Vitamin D Deficiency | interventions — Calcifediol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CTAP101 Capsules 900mcg/weekly (Active Comparator): CTAP101 Oral Capsules/Calcifediol, calcidiol, 25-hydroxyvitamin D3, 900mcg/weekly for 26 weeks
  Interventions: Drug: Calcifediol Oral Capsule
- Placebo Capsules weekly (Placebo Comparator): Placebo Oral Capsules/weekly for 26 weeks
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Calcifediol Oral Capsule — Capsule, weekly
  Other Names: CTAP101
  Arms: CTAP101 Capsules 900mcg/weekly
Drug: Placebo oral capsule — Capsule, weekly
  Arms: Placebo Capsules weekly

SUMMARY:
Safety, Efficacy, PK and PD of CTAP101 (calcifediol) ER Capsules for SHPT in HD Patients VDI

DETAILED DESCRIPTION:
A Multi-Center, Randomized, Two-Cohort Phase 2 Study to Evaluate the Safety, Efficacy, Pharmacokinetics (PK) and Pharmacodynamics (PD) of CTAP101 (calcifediol) Extended-Release Capsules to Treat Secondary Hyperparathyroidism (SHPT) in Subjects with Vitamin D Insufficiency (VDI) and Chronic Kidney Disease Requiring Regular Hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet the following criteria to be enrolled in this study:

1. Be at least 18 years of age.
2. Be diagnosed with CKD requiring in-center HD tiw for the preceding 6 months, as confirmed by medical history.
3. Be without any disease state or physical condition that might impair evaluation of safety or which, in the investigator's opinion, would interfere with study participation, including:

   1. Serum albumin ≤ 3.0 g/dL; and,
   2. Serum transaminase (alanine transaminase [ALT], glutamic pyruvic transaminase [SGPT], aspartate aminotransferase [AST] or glutamic oxaloacetic transaminase [SGOT]) > 2.5 times the upper limit of normal at screening.
4. Be receiving calcimimetic therapy (either etelcalcetide or cinacalcet) and/or calcitriol or other 1α-hydroxylated vitamin D analog (paricalcitol or doxercalciferol) for at least 1 month at the time of screening for enrollment. Approximately 50% of enrolled subjects will have been receiving calcimimetic therapy.
5. Exhibit during the initial screening visit:

   1. Plasma immunoreactive parathyroid hormone (iPTH) ≥150 pg/mL and <600 pg/mL if receiving etelcalcetide, cinacalcet, calcitriol or other 1α-hydroxylated vitamin D analog (paricalcitol or doxercalciferol); or
   2. Plasma iPTH ≥300 pg/mL and <900 pg/mL if not receiving etelcalcetide, cinacalcet, calcitriol or other 1α-hydroxylated vitamin D analog; and,
   3. Serum total 25-hydroxyvitamin D <30 ng/mL if not receiving vitamin D supplementation.
6. When otherwise confirmed eligible at Visit 1, must forgo any further treatment with etelcalcetide and cinacalcet for the duration of the study and undergo an 8-week washout period.
7. When otherwise confirmed eligible at Visit 1, must forgo any further treatment with calcitriol or other 1α-hydroxylated vitamin D analogs or vitamin D supplements for the duration of the study and undergo an 8-week washout period.
8. Exhibit after the 8-week washout period (if required due to prior use of etelcalcetide, cinacalcet, calcitriol or other 1α-hydroxylated vitamin D analogs, or vitamin D supplementation):

   1. Plasma iPTH increased by at least 50%;
   2. Plasma iPTH ≥300 pg/mL and <1,200 pg/mL;
   3. Corrected serum calcium <9.8 mg/dL;
   4. Serum total 25-hydroxyvitamin D <50 ng/mL; and,
   5. Serum phosphorus <6.5 mg/dL.
9. When otherwise confirmed eligible at Visit 1, if taking more than 1,000 mg per day of elemental calcium, reduce calcium use (to ≤1,000 mg per day) and/or use non-calcium based phosphate binder therapies (as needed) for the duration of the study.
10. When otherwise confirmed eligible at Visit 1, if taking bone metabolism therapies that may interfere with study endpoints, must discontinue use of these agents for the duration of the study.
11. Willing and able to comply with study instructions and commit to all clinic visits for the duration of the study.
12. Female subjects of childbearing potential must be neither pregnant nor lactating and must have a negative serum beta-human chorionic gonadotropin (b-hCG) pregnancy test at the first screening visit and at other scheduled times.
13. All female subjects of childbearing potential and male subjects with female partners of childbearing potential must agree to use effective contraception (eg, implants, injectables, combined oral contraceptives, intrauterine device, sexual abstinence, vasectomy or vasectomized partner) for the duration of the study.
14. Be able to read, understand and sign the subject Informed Consent Form (ICF) or have a legal representative sign the ICF.

4.3 Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from the study:

1. Scheduled kidney transplant or parathyroidectomy.
2. History (prior 2 months) of corrected serum calcium ≥9.8 mg/dL or serum phosphorus

   ≥6.5 mg/dL if not receiving calcitriol or other 1α-hydroxylated vitamin D analog.
3. Receipt of bisphosphonate therapy or other bone modifying treatment (eg, denosumab) within 6 months prior to enrollment.
4. Known previous or concomitant serious illness or medical condition, such as malignancy, human immunodeficiency virus, significant gastrointestinal or hepatic disease, intestinal malabsorption disorder, hepatitis or cardiovascular event that in the opinion of the investigator may worsen or reduce life expectancy, and/or interfere with participation in the study.
5. History of neurological/psychiatric disorder, including psychotic disorder or dementia, or any reason which, in the opinion of the investigator makes adherence to a treatment or follow-up schedule unlikely.
6. Known or suspected hypersensitivity to any of the constituents of the study drugs.
7. Currently participating in, or has participated in, an interventional/investigational study within 30 days prior to study screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - AKDHC Medical Research Services, Peoria, Arizona
  - AKDHC Medical Research Services, Phoenix, Arizona
  - WCCT Global, Inc., Cypress, California
  - Hacienda Dialysis Center, Hacienda Heights, California
  - California Institute of Renal Research CKD/Dialysis & Transplant Division, La Mesa, California
  - Long Beach Quest Dialysis Center, Long Beach, California
  - Ontario Dialysis Center, Ontario, California
  - North America Research Institute, Inc., San Dimas, California
  - Laurel Canyon Dialysis, LLC, Sun Valley, California
  - University of Colorado Denver Anschutz Medical Campus, Aurora, Colorado
  - Research by Design, LLC, Chicago, Illinois
  - Northshore University Health, Evanston, Illinois
  - Renal and Transplant Associates of New England, Springfield, Massachusetts
  - Southwest MS Nephrology, McComb, Mississippi
  - Southwest Houston Research LTD, Houston, Texas
  - Kidney & Hypertension Specialists, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CTAP101 Capsules 900mcg/Weekly | Placebo Capsules Weekly
Started | 33 | 11
Completed | 25 | 8
Not Completed | 8 | 3
Not completed — Adverse Event | 5 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Subject moving out of state | 1 | 0

BASELINE CHARACTERISTICS:
Population: Modified intention-to-treat (mITT) population.
Groups:
- Total: Total of all reporting groups
Arm/Group | CTAP101 Capsules 900mcg/Weekly | Placebo Capsules Weekly | Total
Number analyzed (Participants) | 28 | 9 | 37
Age, Customized [Count of Participants; unit: Participants]
  < 65 years old | 21 | 7 | 28
  >= 65 years old | 7 | 2 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 17
  Male | 16 | 4 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 23 | 5 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 5 | 25
  White | 7 | 4 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response During Efficacy Assessment Period
Description: To evaluate the efficacy of repeated dosing with 900 mcg per week of CTAP101 extended release (ER) Capsules versus placebo in raising mean serum total 25-hydroxyvitamin D (25D) to ≥50 ng/mL and in reducing mean plasma intact parathyroid hormone (iPTH) by at least 30% from pre-treatment baseline.
Time Frame: 26 weeks
Population: mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | CTAP101 Capsules 900mcg/Weekly | Placebo Capsules Weekly
Number analyzed (Participants) | 28 | 9
Participants | 4 | 0
Statistical Analysis 1: Comparison: CTAP101 Capsules 900mcg/Weekly vs Placebo Capsules Weekly; Test type: Other; p = 0.5536, Fisher Exact

2. Primary Outcome: Total 25-hydroxyvitamin D Response Analysis During Efficacy Period
Description: Summary of participants with mean serum total 25-hydroxyvitamin D ≥50 ng/mL at the end of treatment
Time Frame: 26 weeks
Population: mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | CTAP101 Capsules 900mcg/Weekly | Placebo Capsules Weekly
Number analyzed (Participants) | 28 | 9
Participants | 28 | 1

3. Primary Outcome: Number of Participants With Intact Parathyroid Hormone (iPTH) Response During Efficacy Assessment Period
Description: Summary of participants who experienced a reduction in mean plasma iPTH by greater than 30% from the pre-treatment baseline
Time Frame: 26 weeks
Population: mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | CTAP101 Capsules 900mcg/Weekly | Placebo Capsules Weekly
Number analyzed (Participants) | 28 | 9
Participants | 4 | 0

4. Primary Outcome: Pharmacokinetic (PK) Profile (Cmax) of Serum Calcifediol
Description: To assess Cmax of serum calcifediol after a single dose of 900 mcg at the start of the study (Single Dose PK Period), and a repeat dose of 300 mcg at the end of the study (Repeat Dose PK Period)
Time Frame: 0, 4, 8, 12, 16, 20, 24, 30, 36, 42 and 48 hours post-dose (single and repeat dose)
Population: PK population. 6 subjects did not complete the repeat PK dosing.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- CTAP101 Capsules 900mcg: PK subgroup
Arm/Group | CTAP101 Capsules 900mcg
Number analyzed (Participants) | 18
ng/mL
  Cmax (single PK) | 45.5 (20.17)
  Cmax (repeat PK): number analyzed (Participants) | 12
  Cmax (repeat PK) | 181.0 (171.92)

5. Primary Outcome: Pharmacokinetic (PK) Profile (Tmax) of Serum Calcifediol
Description: To assess Tmax of serum calcifediol after a single dose of 900 mcg at the start of the study (Single Dose PK Period), and a repeat dose of 300 mcg at the end of the study (Repeat Dose PK Period)
Time Frame: 0, 4, 8, 12, 16, 20, 24, 30, 36, 42 and 48 hours post-dose (single and repeat dose)
Population: PK population. 6 subjects did not complete the repeat PK dosing.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CTAP101 Capsules 900mcg
Number analyzed (Participants) | 18
hours
  Tmax (single PK) | 0.6 (0.41)
  Tmax (repeat PK): number analyzed (Participants) | 12
  Tmax (repeat PK) | 2.5 (2.72)

6. Primary Outcome: Pharmacokinetic (PK) Profile (AUC0-t) of Serum Calcifediol
Description: To assess AUC0-t of serum calcifediol after a single dose of 900 mcg at the start of the study (Single Dose PK Period), and a repeat dose of 300 mcg at the end of the study (Repeat Dose PK Period)
Time Frame: 0, 4, 8, 12, 16, 20, 24, 30, 36, 42 and 48 hours post-dose (single and repeat dose)
Population: PK population. 6 subjects did not complete the repeat PK dosing.
Measure: Mean (Standard Deviation); unit: hour x ng/mL
Arm/Group | CTAP101 Capsules 900mcg
Number analyzed (Participants) | 18
hour x ng/mL
  AUC0-t (single PK) | 9118.4 (3557.65)
  AUC0-t (repeat PK): number analyzed (Participants) | 12
  AUC0-t (repeat PK) | 95820.7 (44858.77)

7. Secondary Outcome: Pharmacodynamic Analysis of 1,25-dihydroxyvitamin D
Description: Effect of CTAP101 on 1,25-dihydroxyvitamin D
Time Frame: 26 weeks
Population: mITT population.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | CTAP101 Capsules 900mcg/Weekly | Placebo Capsules Weekly
Number analyzed (Participants) | 28 | 9
pg/mL
  Baseline | 9.4 (1.2) | 12.6 (2.7)
  Visit 24 | 50.7 (7.8) | 13.4 (4.1)

ADVERSE EVENTS:
Time Frame: 26 weeks
Description: Safety population. CTAP101 group has 32 subjects and placebo group has 11 subjects who received at least 1 dose.
Arm/Group | CTAP101 Capsules 900mcg/Weekly | Placebo Capsules Weekly
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/11
Serious Adverse Events (participants affected / at risk) | 15/32 | 4/11
Other Adverse Events (participants affected / at risk) | 29/32 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CTAP101 Capsules 900mcg/Weekly (N=32) | Placebo Capsules Weekly (N=11)
Corona virus infection (Infections and infestations) | 3 | 1
Osteomyelitis (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 0 | 1
Septic embolus (Infections and infestations) | 2 | 0
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 1
Presyncope (Nervous system disorders) | 2 | 0
Demyelinating polyneuropathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Incision site complication (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CTAP101 Capsules 900mcg/Weekly (N=32) | Placebo Capsules Weekly (N=11)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 1
Cardiomegaly (Cardiac disorders) | 2 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 3 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Eye pain (Eye disorders) | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Gastrointestinal angiectasia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Jejunal ulcer (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Asthenia (General disorders) | 0 | 1
Feeling abnormal (General disorders) | 1 | 0
Feeling hot (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Localised oedema (General disorders) | 1 | 0
Malaise (General disorders) | 3 | 0
Pyrexia (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Infectious colitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Tracheobronchitis viral (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 3 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 3 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2 | 0
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0
Complications of transplant surgery (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 1
Vascular access malfunction (Injury, poisoning and procedural complications) | 3 | 0
Breath sounds abnormal (Investigations) | 1 | 0
Coronavirus test positive (Investigations) | 1 | 1
Intraocular pressure test (Investigations) | 1 | 0
Troponin increased (Investigations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
IIIrd nerve paralysis (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Unresponsive to stimuli (Nervous system disorders) | 1 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Breast oedema (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary vascular disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 1
Hypertensive emergency (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 5 | 3
Peripheral ischaemia (Vascular disorders) | 1 | 0
Steal syndrome (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT03602261/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT03602261/SAP_001.pdf